CLINICAL TRIAL: NCT04688541
Title: A Preliminary Randomised Crossover Study to Determine User Acceptability and Laboratory Data Regarding Use of a Novel Indwelling Urinary Catheter: the Optitip Study
Brief Title: A Study to Determine User Acceptability and Laboratory Data Regarding Use of a Novel Indwelling Urinary Catheter: the Optitip Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Consequence of COVID-19 pandemic all staff working on this study were moved elsewhere and never returned to complete this work. Full RCT 'CADET' looking into Optitip use now taking place, so this pilot work is no longer required.
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ERGO 53798
Record Dates: First submitted 2020-04-21; First posted 2020-12-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-10

CONDITIONS: Urologic Diseases
Keywords: Catheter; Pilot; Biofilm
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First standard Foley catheter than Optitip catheter (Active Comparator): Each participant is given the 2 trial catheters for successive periods of 4 weeks (+ up to 7 days) for each treatment period:
  Study period 1 = Standard Foley catheter Study period 2 = Optitip catheter
  Interventions: Device: Optitip Catheter (LinC Medical); Device: Foley catheter
- First Optitip catheter than standard Foley catheter (Active Comparator): Each participant is given the 2 trial catheters for successive periods of 4 weeks (+ up to 7 days) for each treatment period:
  Study period 1 = Optitip catheter Study period 2 = Standard Foley catheter
  Interventions: Device: Optitip Catheter (LinC Medical); Device: Foley catheter

INTERVENTIONS:
Device: Optitip Catheter (LinC Medical) — The Optitip catheter, unlike the Foley catheter design which has a protruding tip, the Optitip has a blunt open end (eyelet) that protrudes slightly beyond a single fluid-filled 10ml balloon. It has an additional drainage eyelet underneath the balloon.
Device: Foley catheter — Foley catheter

SUMMARY:
In this study, long-term catheter patients in the Community setting (both catheter clinic attenders or home catheter changes) will be invited to participate in a randomised cross-over study to compare their standard Foley catheter with the Optitip catheter. The participants will be randomised to Arm A (Standard Foley catheter then Optitip) or Arm B (Optitip then Standard Foley catheter) and will have each catheter inserted for successive periods of 4 weeks (+ up to 7 days). The catheters will be collected following removal and analysed for presence of biofilm; catheter specimens of urine will also be collected to measure detection/quantity microorganisms and cytokines. The quality of life of participants will be assessed at baseline and the end of each study period using a validated quality of life tool for long-term catheter users - the ICIQ-LTCqol.

DETAILED DESCRIPTION:
When normal bladder emptying is not possible due to injury, disease, surgery, or neurological conditions, an indwelling urinary catheter (IUC) may be required. An estimated 90,000 people in the UK require a long-term urinary catheter.

Urinary catheters are associated with significant harm and can cause substantial distress. Furthermore, managing frequent catheter-associated problems is a resource intensive burden to the providers of community healthcare services Currently, most patients use the standard Foley catheter design and experience problems that can constrain work and social lives, lead to UTI and pain and substantially reduce quality of life.

The Optitip catheter became available on the Drug Tariff in 2017. Unlike the Foley catheter design which has a protruding tip, the Optitip has a blunt open end (eyelet) that protrudes slightly beyond a single fluid-filled 10ml balloon. It has an additional drainage eyelet underneath the balloon.

The Optitip therefore has the potential to make important differences to patients by reducing pain/discomfort; reducing blockage frequency and potentially reducing clinical infection.

ELIGIBILITY:
Inclusion Criteria:

* Existing patients of Solent NHS Trust for > 3months
* Capable of giving informed consent
* Adult men or women (≥18)
* Planning to be using a long-term catheter for the duration of the study (3 months)
* Able to attend the clinic on the clinic/research days for catheter changes or have a research nurse visit them at home to do the changes
* Willing to have the next 2 catheter changes at 4 weekly intervals, which may be different from their usual change interval

Exclusion Criteria:

* Currently pregnant or planning to become pregnant
* Lack of capacity to consent
* Currently taking antibiotics for any reason (not just UTI) - unless the patient is usually on long term prophylactic antibiotics they may continue as long as they do so for the duration of the trial (unless instructed otherwise by a medical professional)
* Taken antibiotics for any reason in the previous month
* Has frequent catheter blockage ie. requiring catheter changes usually less than 4 weekly or visits for other catheter related reasons more frequently than 4 weekly
* Planned bladder washouts of any frequency
* Suprapubic catheter users
* Those who need to visit a urology clinic due to complex catheter changes
* Participation in a related study
* Using a non-standard catheter e.g. not a Foley design
* Using an unusual sized catheter - outside the sizes available (12-18F)
* Unable to complete the assessments in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of blockage - accumulation of biofilm | 4 weeks + up to 7 days.
  To compare the accumulation of biofilm on the catheter surface as a marker for the likelihood of blockage following 4 weeks insertion of an Optitip catheter to 4 weeks insertion of a standard Foley catheter. The 2 catheters (Foley and Optitip) will be collected and sent to the laboratory immediately after removal - the insertion period is 4 weeks + up to 7 days.

SECONDARY OUTCOMES:
Participant completion of the validated quality of life tool - ICIQ-LTCqol. | 56 days (+ up to 14 days)
  To determine whether there is any difference in patient reported quality of life score after using an Optitip catheter compared with a standard Foley catheter. Catheter function and concern 0-42 score, Lifestyle impact 0-15. Higher score better quality of life.
Quantify microorganisms in the urine. | 56 days (+ up to 14 days)
  Analysis of CSU for micro-organisms. To determine whether there is any difference in micro-organism in urine samples collected following the use of an Optitip catheter compared to a standard Foley catheter.
Quantify cytokines in the urine. | 56 days (+ up to 14 days)
  Analysis of CSU for cytokines. To determine whether there is any difference in cytokines in urine samples collected following the use of an Optitip catheter compared to a standard Foley catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Fader, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: No
At all times throughout the study, confidentiality will be observed by all parties. All data shall be secured against unauthorised access whilst privacy and confidentiality of information about each participant shall be preserved in reports and any publication. Each participant will be assigned a unique identification number at the time of enrolment.
  The investigator will maintain a confidential study enrolment list. This will contain the unique assigned identification number and name. The investigator bears the responsibility of keeping this list confidential.